CLINICAL TRIAL: NCT07347717
Title: A Digital Self-Compassion Writing Intervention to Improve the Mental Health of Parents of Autistic Individuals
Brief Title: Digital Self-Compassion Writing Intervention to Support Mental Health of Parents of Autistic Individuals
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Macau (Other)
Responsible Party: Principal Investigator, Peilian Chi, Associate Professor, University of Macau
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MYRG-GRG2024-00269-FSS
Record Dates: First submitted 2025-12-22; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Mental Health
Keywords: Digital self-compassion writing intervention
MeSH Terms: conditions — Psychological Well-Being | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-compassion writing group (Experimental): This digital intervention is a 14-day writing program delivered via a WeChat mini-program. Each day, participants complete a two-step writing task: (1) mindfully describe an event and their feelings, and (2) support themselves with self-kindness. Daily reminders are sent to encourage engagement. Each session takes approximately 5 minutes. The program is tailored for parents of autistic individuals to provide a brief, low-cost mental health support option for chronically stressed caregivers.
  Interventions: Behavioral: Self-compassion writing group
- Control group (Active Comparator): Participants in the control group use the same mini-program for 14 days but complete factual writing tasks. They are instructed to recall their day and describe events objectively, without emotional content or cognitive reframing. This controls for time, attention, and writing activity.
  Interventions: Behavioral: Control group (placebo)

INTERVENTIONS:
Behavioral: Self-compassion writing group — This digital intervention is a 14-day writing program delivered via a WeChat mini-program. Each day, participants complete a two-step writing task: (1) mindfully describe an event and their feelings, and (2) support themselves with self-kindness. Daily reminders are sent to encourage engagement. Each session takes approximately 5 minutes. The program is tailored for parents of autistic individuals to provide a brief, low-cost mental health support option for chronically stressed caregivers.
  Arms: Self-compassion writing group
Behavioral: Control group (placebo) — Participants in the control group use the same mini-program for 14 days but complete factual writing tasks. They are instructed to recall their day and describe events objectively, without emotional content or cognitive reframing. This controls for time, attention, and writing activity.
  Arms: Control group

SUMMARY:
This randomized controlled trial aims to evaluate the feasibility, acceptability, and preliminary efficacy of a digital self-compassion writing intervention for parents of autistic individuals. Participants will engage in a 14-day self-compassion writing program delivered via a WeChat mini-program. The study seeks to answer the following questions:

* Is the study design and digital self-compassion writing intervention feasible and acceptable for parents of autistic individuals?
* Does the intervention lead to greater improvements in self-compassion and mental health outcomes compared to the control group?
* Do baseline characteristics moderate the intervention effect compared to the control group?
* Among intervention participants, do satisfaction and usage patterns predict greater improvements in outcomes?
* Does improvement in self-compassion mediate changes in mental health outcomes?

ELIGIBILITY:
Inclusion Criteria:

* are parents of individuals with either a formal autism diagnosis or a provisional diagnosis from a medical institution
* are living with the autistic individual
* are aged 18 years or older
* regularly use WeChat
* are willing to commit to the study procedure

Exclusion Criteria:

* current experience of acute mental health issues (e.g., severe depression, anxiety, suicidal tendencies)
* undergoing serious health crises (e.g., undergoing major surgery or diagnosed with a life-threatening illness)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
Eligibility rate | From date of initial registration until eligibility determination, typically within 2 days of registration (up to 10 days maximum)
  Proportion of registrants who met all inclusion criteria (n_eligible / n_registered). This metric evaluates the effectiveness of the registration form in screening for eligibility.
Baseline questionnaire completion rate | From date of eligibility confirmation until completion of baseline assessment, up to 10 days maximum
  Proportion of eligible registrants who completed the baseline assessment (n_baseline / n_eligible)
Post-intervention questionnaire completion rate | From date of completion of baseline assessment until completion of post-intervention assessment, typically within 1 day after intervention (up to 2 days maximum)
  Proportion of baseline completers who complete the post-intervention questionnaire (n_post / n_baseline)
Follow-up questionnaire completion rate | From date of completion of the post-intervention assessment until 14 days after completion of the follow-up assessment (up to 15 days maximum).
  Proportion of post-intervention assessment completers who provided follow-up data (n_follow / n_post).
Intervention satisfaction | Measured at the post-intervention assessment, conducted within two days after the end of the intervention
  A 4-item measure assessing satisfaction with the intervention. Items are rated on a 5-point Likert scale. Total scores are obtained by averaging item scores. Higher scores indicate higher satisfaction with the intervention.
Intervention adherence | During the 14-day intervention period.
  Measured by the average number of entries submitted during the intervention period.
Intervention fidelity | During the 14-day intervention period.
  Measured by the proportion of entries that meet the criteria for intervention and control groups, respectively. Evaluated after intervention completion by reviewing all entries submitted during the 14-day intervention period.
Self-compassion | Measured at three time points: baseline (prior to intervention), immediately post-intervention (within 2 days after intervention ends), and at two-week follow-up (15-16 days after intervention completion).
  A 13-item measure (positive subscale of the Self-Compassion Scale) assessing self-compassion across three components: mindfulness, common humanity, and self-kindness. Items are rated on a 5-point Likert scale (1 = almost never, 5 = almost always). Total and subscale scores are calculated by averaging item responses. Higher scores indicate greater self-compassion.

SECONDARY OUTCOMES:
Emotion regulation | Measured at three time points: baseline (prior to intervention), immediately post-intervention (within 2 days after intervention ends), and at two-week follow-up (15-16 days after intervention completion).
  A six-item scale (Emotion Regulation Questionnaire-Short Form, ERQ-S) measuring two emotion regulation strategies: cognitive reappraisal and expression suppression. Items are rated on a 7-point Likert scale. Subscale scores are calculated by summing item scores within each strategy. Higher scores indicate more frequent use of that emotion regulation strategy.
Psychological flexibility | Measured at three time points: baseline (prior to intervention), immediately post-intervention (within 2 days after intervention ends), and at two-week follow-up (15-16 days after intervention completion).
  A six-item scale (Psy-Flex) measuring psychological flexibility. Items are rated on a 7-point Likert scale. Total scores are calculated by summing item scores. Higher scores indicate higher levels of psychological flexibility.
Well-being | Measured at three time points: baseline (prior to intervention), immediately post-intervention (within 2 days after intervention ends), and at two-week follow-up (15-16 days after intervention completion).
  5 items (WHO Well-Being Index, WHO-5). Total scores are calculated by summing item scores, ranging from 0 to 25. Higher scores indicate higher levels of well-being.
Flourishing | Measured at three time points: baseline (prior to intervention), immediately post-intervention (within 2 days after intervention ends), and at two-week follow-up (15-16 days after intervention completion).
  8 items (Flourishing Scale). Total scores are calculated by averaging item scores, ranging from 1 to 7. Higher scores indicate higher levels of flourishing.
Life satisfaction | Measured at three time points: baseline (prior to intervention), immediately post-intervention (within 2 days after intervention ends), and at two-week follow-up (15-16 days after intervention completion).
  A single-item measuring life satisfaction rated on a 0-10 reponse scale (0 = not at all, 10 = completely).
Stress | Measured at three time points: baseline (prior to intervention), immediately post-intervention (within 2 days after intervention ends), and at two-week follow-up (15-16 days after intervention completion).
  Stress will be measured by the single-item subjective level of stress (SLS-1). 0 = not at all, 5 = moderate, 10 = extremely.
Anxiety | Measured at three time points: baseline (prior to intervention), immediately post-intervention (within 2 days after intervention ends), and at two-week follow-up (15-16 days after intervention completion).
  7 items (Generalized Anxiety Disorder-7, GAD-7). Total scores range from 0 to 21, with higher scores indicating higher levels of anxiety.
Depression | Measured at three time points: baseline (prior to intervention), immediately post-intervention (within 2 days after intervention ends), and at two-week follow-up (15-16 days after intervention completion).
  9 items (Patient Health Questionnaire-9, PHQ-9). Total scores range from 0 to 27, with higher scores indicating higher levels of depression.
Sleep quality | Measured at three time points: baseline (prior to intervention), immediately post-intervention (within 2 days after intervention ends), and at two-week follow-up (15-16 days after intervention completion).
  1 item (Single-Item Sleep Quality Scale). Possible ratings range from 0 to 10, with higher ratings indicating better sleep quality.
Parenting stress | Measured at three time points: baseline (prior to intervention), immediately post-intervention (within 2 days after intervention ends), and at two-week follow-up (15-16 days after intervention completion).
  15 items (Simplified Parenting Stress Index/Short Form-15, S-PSI/SF). Total scores are calculated by summing item scores, ranging from 15 to 75. Higher scores indicate higher levels of parenting stress.
Parenting efficacy | Measured at three time points: baseline (prior to intervention), immediately post-intervention (within 2 days after intervention ends), and at two-week follow-up (15-16 days after intervention completion).
  4 items (Me as a Parent Scale-Short Form). Total scores are calculated by summing item scores, ranging from 4 to 20. Higher scores indicate higher levels of parenting efficacy.
Parenting practices | Measured at three time points: baseline (prior to intervention), immediately post-intervention (within 2 days after intervention ends), and at two-week follow-up (15-16 days after intervention completion).
  27 items (Multidimensional Assessment of Parenting Scale) that reflect positive and negative parenting practices are used. Scores for positive parenting and negative parenting will be calculated by summing item scores, respectively.
Child adjustment | Measured at three time points: baseline (prior to intervention), immediately post-intervention (within 2 days after intervention ends), and at two-week follow-up (15-16 days after intervention completion).
  24 items (Child Adjustment and Parent Efficacy Scale-Developmental Disability, CAPES-DD). To obtain a Behavioral Problems subscale score, sum ratings for items 1, 3, 4, 5, 6, 7, 8, 9, 10, and 12, with a possible range from 0 to 30. To obtain an Emotional Problems subscale score, sum ratings for items 2, 11, and 13 with a possible range from 0 to 9. Higher scores indicate greater levels of child emotional or behavioral problems. To obtain a Prosocial Behavior scale score, sum ratings for items 17, 18, 19, 20, 21, 22, 23, and 24, with a possible range from 0 to 24.
Daily self-compassion | Daily during the 14-day intervention period
  A 3-item measure assessing self-compassion components (mindfulness, common humanity, and self-kindness) immediately after each writing session. Items are rated on a 5-point Likert scale. Higher scores indicate greater self-compassion.
Daily positive affect | Daily during the 14-day intervention period.
  A single-item measure assessing positive emotions immediately after each writing session. This item is rated on a 5-point Likert scale. Higher scores indicate greater positive emotions.
Daily life satisfaction | Daily during the 14-day intervention period
  A single-item measure assessing life satisfaction immediately after each writing session. This item is rated on a 5-point Likert scale. Higher scores indicate greater life satisfaction.
Daily parenting efficacy | Daily during the 14-day intervention period
  A single-item measure assessing parenting efficacy immediately after each writing session. This item is rated on a 5-point Likert scale. Higher scores indicate greater parenting efficacy.

OTHER OUTCOMES:
Personality | Measured at three time points: baseline (prior to intervention), immediately post-intervention (within 2 days after intervention ends), and at two-week follow-up (15-16 days after intervention completion).
  Will be measured by the Ten-Item Personality Inventory in Chinese. Scale scoring ("R" denotes reverse-scored items): Extraversion: 1, 6R; Agreeableness: 2R, 7; Conscientiousness: 3, 8R; Emotional Stability: 4R, 9; Openness to Experiences: 5, 10R.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Macau, Taipa, Macau

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Analytic Code
Time Frame: The IPD and supporting information will be made available after the publication of study results, anticipated around December 2027. There will be no specified end date for availability.
Access Criteria: The IPD and supporting information will be available upon reasonable request to the corresponding author. Researchers or qualified professionals may request access to de-identified data and analytic code for purposes such as secondary analysis or replication. Requests will be reviewed to ensure appropriate use and data protection.